CLINICAL TRIAL: NCT02818686
Title: A Phase 1b Multi-Center, Randomized, Double-Blind, Multi-Dose, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Plasma Exposure of TD-1473 in Subjects With Moderately-to-Severely Active Ulcerative Colitis
Brief Title: TD-1473 for Active Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0144; 2016-001633-27 (EudraCT Number)
Record Dates: First submitted 2016-06-23; First posted 2016-06-30 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis, Active Moderate; Ulcerative Colitis, Active Severe
Keywords: Ulcerative Colitis, Active Moderate and Severe
MeSH Terms: conditions — Colitis, Ulcerative | interventions — izencitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TD-1473 low dose (Experimental): 10 subjects will be randomized to receive low-dose TD-1473 orally daily for 28 days
  Interventions: Drug: TD-1473
- TD-1473 mid dose (Experimental): 10 subjects will be randomized to receive mid-dose TD-1473 orally daily for 28 days
  Interventions: Drug: TD-1473
- TD-1473 high dose (Experimental): 10 subjects will be randomized to receive high-dose TD-1473 orally daily for 28 days
  Interventions: Drug: TD-1473
- Placebo (Placebo Comparator): 10 subjects will be randomized to receive placebo orally daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1473
  Arms: TD-1473 high dose; TD-1473 low dose; TD-1473 mid dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of TD-1473 in subjects with moderately-to-severely active UC over 28 days. This exploratory study will also serve as a signal seeking endeavor to demonstrate biologic effect associated with TD-1473 through biomarker analysis and clinical, endoscopic, and histologic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Has a history of ulcerative colitis diagnosis at least 3 months prior to screening
* Is intolerant, refractory, or only partially responsive to aminosalicylates, corticosteroids, immunomodulators, or biologics. If subject is currently receiving an oral aminosalicylate, he or she is eligible and can stay on that dose of aminosalicylate provided the dose has been stable for at least 2 weeks prior to screening. If the subject is currently receiving an oral corticosteroid, he or she is eligible if the dose is equivalent to or less than prednisone 20 mg/day or budesonide 9 mg/day and stable for at least 2 weeks prior to screening sigmoidoscopy if the subject has been on corticosteroids for more than 2 weeks.
* Has a rectal bleeding score ≥ 1 and a bowel frequency score ≥ 1 on the patient-reported outcome 2 (PRO2) on screening sigmoidoscopy day and on Day 1 in addition to a modified Mayo endoscopic subscore of ≥ 2 during screening
* Women of childbearing potential must have a negative pregnancy test and either abstain from sexual intercourse or use a highly effective method of birth control
* Willing and able to give informed consent
* Additional inclusion criteria apply

Exclusion Criteria:

* Has fulminant colitis, toxic megacolon, primary sclerosing cholangitis, Crohn's disease, history of colitis-associated colonic dysplasia, active peptic ulcer disease
* Medications of exclusion: a) azathioprine, 6-mercaptopurine, or methotrexate within the 28 days prior to Day 1, b) adalimumab, infliximab, golimumab, etanercept, or certolizumab within the 60 days prior to Day 1, c) intravenous corticosteroids within the 14 days prior to Day 1, d) topical mesalamine or steroid (i.e., enemas or suppositories) within the 14 days prior to Day 1, e) any prior exposure to mycophenolic acid, tacrolimus, sirolimus, cyclosporine, natalizumab, rituximab, efalizumab, ustekinumab, fingolimod, or thalidomide, f) NSAIDs on a daily basis, g) tofacitinib within the 60 days prior to Day 1; h) vedolizumab within 120 days prior to Day 1
* Has a current bacterial, parasitic, fungal, or viral infection
* Is positive for hepatitis A, B or C, HIV or tuberculosis
* Has clinically significant abnormalities in laboratory evaluations
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to screening (or within 60 days prior to screening if investigational drug was a biologic or another Janus kinase (JAK) inhibitor, or is currently participating in another trial of an investigational drug (or medical device)
* Use of prescription medications started or with a dose adjustment within 4 weeks prior to study enrollment, or over-the-counter medications or supplements started or with a dose adjustment within 2 weeks prior study enrollment. Anti-diarrheal medications are allowed only if dose has been stable at least 2 weeks prior to study enrollment
* Additional exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events (TEAE) | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experience one or more treatment-emergent Adverse Events (TEAE)
Moderate or Severe Treatment-emergent Adverse Events (TEAE) | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experience one or more moderate or severe treatment-emergent Adverse Events (TEAE)
Serious Treatment-emergent Adverse Events (TEAE) | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experience one or more serious treatment-emergent Adverse Events (TEAE)
Clinical Laboratory Measurements | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experienced a Clinically Significant Clinical Laboratory Measurements
Electrocardiogram | Baseline to Day 14
  Number of participants who experienced a Clinically Significant Electrocardiogram (ECG) Result
Vital Signs | Baseline to end of follow-up (a maximum of 42 days)
  Number of participants who experienced a Clinically Significant Vital Sign Measurement
Cmax in plasma | Day 1 and Day 14
  Maximum Observed Plasma Concentration of TD-1473
Tmax in plasma | Day 1 and Day 14
  Time to Reach Maximum Observed Plasma Concentration (Cmax) of TD-1473
Tlast in plasma | Day 1 and Day 14
  Time to Last Quantifiable Concentration of TD-1473
Ctrough in plasma | Day 14 (Pre-dose)
  Trough Concentration of TD-1473
AUC0-4 in plasma | Day 1 and Day 14
  Area Under the Concentration-time Curve from Time Zero to 4 hours Post-Dose of TD-1473
Ctissue in plasma | Day 28
  Tissue Concentration of TD-1473

SECONDARY OUTCOMES:
C-reactive protein (CRP) | Baseline, Day 14 and Day 28
  Mean Change in Serum C-reactive Protein (CRP)
Fecal Calprotectin | Baseline and Day 28
  Mean Change in Fecal Calprotectin
Partial Mayo score | Baseline, Day 14 and Day 28
  Mean Change in Partial Mayo Score

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (8):
- United States (5):
  - Theravance Biopharma Investigational Site, Scottsdale, Arizona
  - Theravance Biopharma Investigational Site, Monroe, Louisiana
  - Theravance Biopharma Investigational Site, Hermitage, Tennessee
  - Theravance Biopharma Investigational Site, Houston, Texas
  - Theravance Biopharma Investigational Site, San Antonio, Texas
- Theravance Biopharma Investigational Site, Tbilisi, Georgia
- Theravance Biopharma Investigational Site, Chisinau, Moldova
- Theravance Biopharma Investigational Site, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

REFERENCES:
- [Derived] Sandborn WJ, Nguyen DD, Beattie DT, Brassil P, Krey W, Woo J, Situ E, Sana R, Sandvik E, Pulido-Rios MT, Bhandari R, Leighton JA, Ganeshappa R, Boyle DL, Abhyankar B, Kleinschek MA, Graham RA, Panes J. Development of Gut-Selective Pan-Janus Kinase Inhibitor TD-1473 for Ulcerative Colitis: A Translational Medicine Programme. J Crohns Colitis. 2020 Sep 16;14(9):1202-1213. doi: 10.1093/ecco-jcc/jjaa049. PMID 32161949